CLINICAL TRIAL: NCT01439581
Title: Utility of Interface Pressure Mapping
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Wellsense USA Inc. (Industry)
Responsible Party: Principal Investigator, Rob Behrendt, MICU Unit Educator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Interface Pressure Mapping
Record Dates: First submitted 2011-09-22; First posted 2011-09-23 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Ulcers; Bedsores
Keywords: patients; susceptible to; hospital; acquired pressure
MeSH Terms: conditions — Ulcer; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Patients were assigned randomly to either a medical intensive care unit with pressure mapping beds or a unit that did not have them
Oversight: Data Monitoring Committee: No

ARMS (2):
- Patients on mapping systems (Experimental)
  Interventions: Device: Mapping System
- Patients not on mapping systems (Active Comparator)
  Interventions: Device: Non-Mapping System

INTERVENTIONS:
Device: Mapping System — Pressure Sensing coverlet on ICU bed and provides real time feedback to assist in effective patient repositioning
  Arms: Patients on mapping systems
Device: Non-Mapping System — Standard ICU bed with no mapping system
  Arms: Patients not on mapping systems

SUMMARY:
To determine if a device that measures and displays pressure that the patients feel when in bed can help nurses reposition the patient effectively and thereby reduce bedsores in the intensive care unit.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older,
* care giver trained on mapping system

Exclusion Criteria:

* Less than 18 years,
* pregnant women,
* weight greater 550 lbs, and subjects requiring a specialty mattress

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 428 (Actual)
Dates: Start 2011-08; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients Not on Mapping Systems: Mapping System: Pressure Sensing coverlet on ICU bed and provides real time feedback to assist in effective patient repositioning
Period: Overall Study
Arm/Group | Patients on Mapping Systems | Patients Not on Mapping Systems
Started | 216 | 212
Completed | 216 | 212
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients on Mapping Systems | Patients Not on Mapping Systems | Total
Number analyzed (Participants) | 216 | 212 | 428
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 143 | 138 | 281
  >=65 years | 73 | 74 | 147
Age, Continuous [Mean (Full Range); unit: years] | 58.7 [19 to 96] | 56.9 [18 to 93] | 57.8 [18 to 96]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110 | 102 | 212
  Male | 106 | 110 | 216
Region of Enrollment [Number; unit: participants]
  United States | 216 | 212 | 428

OUTCOME MEASURES:

1. Primary Outcome: Pressure Mapping Reducing Hospital Acquired Pressure Ulcers
Description: Comparing number of pressure ulcers when using pressure mapping compared to when not.
Time Frame: Time admitted in the Medical Intensive Care Unit
Measure: Count of Participants; unit: Participants
Arm/Group | Patients on Mapping Systems | Patients Not on Mapping Systems
Number analyzed (Participants) | 216 | 212
Participants | 2 | 10

ADVERSE EVENTS:
Arm/Group | Patients on Mapping Systems | Patients Not on Mapping Systems
Serious Adverse Events (participants affected / at risk) | 0/213 | 0/209
Other Adverse Events (participants affected / at risk) | 0/213 | 0/209

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No